CLINICAL TRIAL: NCT01604993
Title: Acute Effect of Nitrate Supplementation From Natural Dietary Sources on Arterial Stiffness and Aortic and Brachial Blood Pressures: a Double-blind, Placebo-controlled, Randomized, Crossover Clinical Trial in Healthy Adults
Brief Title: Acute Effect of Nitrate From Natural Dietary Sources on Arterial Stiffness and Blood Pressures in Healthy Individuals
Acronym: DNAB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 11216
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: Dietary Nitrates; Arterial Stiffness; Vascular; Blood pressure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- High nitrate dietary source (Experimental): 556 grams of high nitrate spinach soup that is orally consumed as a single dose for 7 days.
  Interventions: Other: Spinach soup
- No Nitrate dietary source (Placebo Comparator): 556g low nitrate asparagus soup; orally consumed as a single does for 7 days.
  Interventions: Other: Asparagus soup

INTERVENTIONS:
Other: Spinach soup — 556 g of high Nitrate spinach soup that is orally consumed as a single dose for 7 days
  Arms: High nitrate dietary source
Other: Asparagus soup — 556 grams of low nitrate asparagus soup that is orally consumed for a period of 7 days as a single does
  Arms: No Nitrate dietary source

SUMMARY:
The purpose of this study is to evaluate the acute effect of a meal high in dietary nitrates on aortic augmentation index, brachial and aortic blood pressures, and subendocardial viability ration (SEVR).

DETAILED DESCRIPTION:
Hypertension has become a common medical condition worldwide, raising public concern regarding the accompanying increase in cardiovascular disease risk and other health risks. Targets for optimal blood pressure are often unmet by conventional pharmaceutical therapies; consequently, complementary and alternative medicines are increasing in popularity among patients wishing to better manage their BP. In the case of hypertension, endothelial dysfunction and cardiovascular disease, a decline in the ability of blood vessels to dilate in response to shear stress is a major contributor to vascular pathology. At the core of these conditions is a decreased ability to synthesize nitric oxide, a potent vasodilatory agent. The proposed study will examine whether or not increasing the intake of dietary nitrate, which can be converted to nitric oxide endogenously, can improve three indices of vascular function that are validated risk factors for CVD: arterial stiffness, as measured by aortic augmentation index (AIx), aortic BP and brachial BP.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 18-50
* Must consider themselves to be in good overall health and be free of any conditions or illnesses Women must be post-menopausal or not pregnant.
* Body mass index (BMI) must be <30kg/m^2.
* Normotensive, as defined by brachial SBP <140mmHg and DBP <90mmHg
* Subjects must also be willing to stop using mouthwash for the duration of their participation in the study.

Exclusion Criteria:

* Women of childbearing age may not be pregnant, planning to become pregnant, or breastfeeding at the time of the study
* BMI >30kg/m^2
* Hypertensive as defined by brachial SBP >140mmHg and/or DBP >90mmHg
* Allergy or sensitivity to the study product, reference therapy or nitrates
* Having any gastrointestinal complication or condition
* Chronic use of medications such as prescription NSAIDs, antacids, blood-thinners, hypertensive medications, medications affecting NO synthesis such as Viagra, and use of antibiotics within one month of the study start
* Individuals who are involved in another clinical trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2011-10; Primary Completion 2012-11 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Aortic augmentation index (arterial stiffness) | At each treatment visits, this measurement will be taken in at baseline, 1, 2, and 3 hours post-treatment.

SECONDARY OUTCOMES:
Peripheral (brachial) and central (aortic) systolic and diastolic blood pressure | Brachial blood pressure will be measured at 0 , 1, 2, and 3 hours post -treatmentbaseline and at 1, 2 and 3 hours at every visit.
Subendocardial viability ratio (SEVR) | At 1 hours intervals starting from baseline and ending at 3 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Vuksan, PhD, Principal Investigator — Risk Factor Modification Centre - St. Michael's Hospital
Locations (1):
- Risk Factor Modification Centre, Toronto, Ontario, Canada